CLINICAL TRIAL: NCT04397354
Title: Intracochlear Dexamethasone Application During Cochlear Implantation for Preserving Cochlear Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof.Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-06

CONDITIONS: Hearing Loss, Sensorineural
Keywords: cochlear implant; dexamethasone
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Injection, Intratympanic

STUDY DESIGN:
Intervention Model Description: Prospective, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): intracochlear dexamethasone application during cochlear implantation
  Interventions: Drug: Intracochlear Dexamethasone
- Group 2 (Active Comparator): intratympanic dexamethasone application during cochlear implantation
  Interventions: Drug: Intratympanic Dexamethasone
- Group 3 (Sham Comparator): No drugs during cochlear implantation
  Interventions: Drug: No additional drugs(control Group)

INTERVENTIONS:
Drug: Intracochlear Dexamethasone — intracochlear injection of dexamethasone with cochlear implantation
  Other Names: intracochlear
  Arms: Group 1
Drug: Intratympanic Dexamethasone — intratympanic injection of dexamethasone with cochlear implantation
  Other Names: intratympanic
  Arms: Group 2
Drug: No additional drugs(control Group) — Control group: No drugs will be injected middle ear with cochlear implantation
  Other Names: No drugs
  Arms: Group 3

SUMMARY:
The protection of cochlear cells is one of the main concerns of cochlear implant surgery. New electrode designs or additional molecules have been used for this purpose. The aim of the study is to test the effect of dexamethasone in two different application methods.

DETAILED DESCRIPTION:
The protection of cochlear cells is one of the main concerns of cochlear implant surgery. New electrode designs or additional molecules have been used for this purpose. The aim of the study is to test the effect of dexamethasone in two different application methods. Participants who will have cochlear implant surgery will be divided into three groups. Group 1 will have intracochlear dexamethasone after the incision of the round window membrane. Group 2 will have intratympanic dexamethasone after the incision of the round window membrane. Group 3 will serve as a control group. All participants will be tested after a week, a month, 3, and 6 months. Impedance and threshold measurements will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sensorineural hearing loss
* Patients who will have cochlear implant surgery with CI422 electrode

Exclusion Criteria:

* Patients with cochlear abnormality
* Patients with auditory neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Electrode Impedance(Ohm) | 1-3 months
  All intra-operative impedance values will be acquired after surgery. They will be repeated in first and 3 rd months
Electrode thresholds(CL) | 1-3 months
  All intra-operative thresholds will be acquired after surgery. They will be repeated in first and 3 rd months

CONTACTS AND LOCATIONS:
Overall Officials: Fazil N Ardic, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The metadata will be shared by a public depository.